CLINICAL TRIAL: NCT01860690
Title: BHCG Level in Day 4,7, in Comparison to Day 10 as an Indicator for Treatment Success
Acronym: BHCG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCG1
Record Dates: First submitted 2012-11-20; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2012-12

CONDITIONS: Ectopic Pregnancy
Keywords: MTX; Ectopic pregnancy; medical treatment
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MTX , treatment outcome (Experimental): patient receiving MTX. in a dosage of 50 mg/m^2 , IM , in single dose
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — 50 mg / meter squer Intramuscular (IM) MTX.

SUMMARY:
The investigators want to compeer BHCG levels after Methotrexate ( MTX). treatment for Ectopic pregnancy in days 4 and 7 after MTX. to day 10 . The hypothesis is that "BHCG" level in day 10 is the best indicator for treatment success , superior to day 4 and 7 . According to the investigators impression BHCG level rises in days 4 and 7 due to destruction of the trophoblast tissue , and only day 10 is an indicator for treatment success

ELIGIBILITY:
Inclusion Criteria:

* patients with ectopic pregnancy
* healthy
* hemodynamic stable
* first ectopic

Exclusion Criteria:

* hemodynamic non-stable
* abnormal liver or kidney function
* allergy reaction to MTX

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
To measure the change of levels of "BHCG" in patients receiving Methotrexate for treatment of ectopic pregnancy in days 4, 7, and 10 post treatment | the change of levels in days 4, 7, and 10 post MTX injection
  To compeer levels of BHCG in days 4 and 7 to day 10 after injection of MTX. for Ectopic pregnancy treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Zvi Klein, Kfar Saba, Israel